CLINICAL TRIAL: NCT00509717
Title: Implementation of a Pharmacy-Intervention to Enhance Prescription and Use of Lipid-Lowering Drugs. A Randomized Trial.
Brief Title: Implementation of a Pharmacy-Intervention to Enhance Prescription and Use of Lipid-Lowering Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Zorgverzekeraar CZ (Other); Scientific Institute for Dutch Pharmacists, The Netherlands (Other)
Responsible Party: Caroline van de Steeg-van Gompel, Scientific Institute for Quality of Healthcare
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: WOK/WINAp/CZ-02
Record Dates: First submitted 2007-02-28; First posted 2007-07-31 (Estimated); Last update posted 2008-07-10 (Estimated); Status verified 2008-07

CONDITIONS: Cardiovascular Diseases
Keywords: quality of health care; prescriptions, drug; anticholesteremic agents; community pharmacy services
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- experimental (Experimental)
  Interventions: Other: intensive implementation programme
- control (Active Comparator)
  Interventions: Other: control

INTERVENTIONS:
Other: intensive implementation programme — educational manual; interactive educational meeting tailored to individual needs; reminders and feedback by 3 newsletters and at least 3 telephone calls.
  Arms: experimental
Other: control — educational manual
  Arms: control

SUMMARY:
The purpose of this study is to determine the effectiveness of maximal support of community pharmacies to implement a pharmaceutical care model for improving underprescription and treatment persistence regarding lipid-lowering medication in patients with cardiovascular disease.

DETAILED DESCRIPTION:
Cardiovascular disease is the main cause of death in large parts of the world. Next to life style changes, pharmaceutical treatment is a keystone in the treatment of cardiovascular disease. Despite the strong evidence for the effectiveness of lipid-lowering therapy, less than half of the people eligible are treated. With specific medication searches in the community pharmacy database, an easy tool for detecting patients who are undertreated is available. Based on this tool, a pharmaceutical care model for improving underprescription and treatment persistence regarding lipid-lowering medication in patients with cardiovascular disease was constructed.

Moreover, it is not known yet how to implement this pharmaceutical care model in community pharmacies effectively. With multifaceted interventions the behaviour of health professionals can be changed. In this study the effectiveness of a maximal support strategy, including interactive educational meetings, reminders, audit and feedback, is compared to a minimal implementation strategy.

ELIGIBILITY:
Inclusion Criteria:

* pharmacies: resident in the south of the Netherlands
* patients: with antiplatelet therapy and without lipid-lowering medication

Exclusion Criteria:for patients:

* terminal disease
* severe mental disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-10; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
The percentage of selected (=undertreated) patients receiving at least one prescription for lipid-lowering medication. | six months after the general practitioner received the list with selected patients

SECONDARY OUTCOMES:
Differences in prescribing for age categories and co-medication. | six months

CONTACTS AND LOCATIONS:
Overall Officials: Peter G. de Smet, PhD, Principal Investigator — Radboud University Medical Center; Michel Wensing, PhD, Study Director — Scientific Institute for Quality of Healthcare
Locations (1):
- UMC St Radboud, Scientific Institute for Quality of Healthcare, Nijmegen, NL, Netherlands

REFERENCES:
- [Background] Mantel-Teeuwisse AK, Verschuren WM, Klungel OH, de Boer A, Kromhout D. Recent trends in (under)treatment of hypercholesterolaemia in the Netherlands. Br J Clin Pharmacol. 2004 Sep;58(3):310-6. doi: 10.1111/j.1365-2125.2004.02152.x. PMID 15327591
- [Background] Blenkinsopp A, Anderson C, Armstrong M. Systematic review of the effectiveness of community pharmacy-based interventions to reduce risk behaviours and risk factors for coronary heart disease. J Public Health Med. 2003 Jun;25(2):144-53. doi: 10.1093/pubmed/fdg030. PMID 12848404
- [Background] Grimshaw JM, Thomas RE, MacLennan G, Fraser C, Ramsay CR, Vale L, Whitty P, Eccles MP, Matowe L, Shirran L, Wensing M, Dijkstra R, Donaldson C. Effectiveness and efficiency of guideline dissemination and implementation strategies. Health Technol Assess. 2004 Feb;8(6):iii-iv, 1-72. doi: 10.3310/hta8060. PMID 14960256
- [Background] Heart Protection Study Collaborative Group. MRC/BHF Heart Protection Study of cholesterol lowering with simvastatin in 20,536 high-risk individuals: a randomised placebo-controlled trial. Lancet. 2002 Jul 6;360(9326):7-22. doi: 10.1016/S0140-6736(02)09327-3. PMID 12114036
- [Background] Gaw A. The care gap: underuse of statin therapy in the elderly. Int J Clin Pract. 2004 Aug;58(8):777-85. doi: 10.1111/j.1368-5031.2004.00300.x. PMID 15372851
- [Background] Teeling M, Bennett K, Feely J. The influence of guidelines on the use of statins: analysis of prescribing trends 1998-2002. Br J Clin Pharmacol. 2005 Feb;59(2):227-32. doi: 10.1111/j.1365-2125.2004.02256.x. PMID 15676046
- [Background] van Wyk JT, Picelli G, Dieleman JP, Mozaffari E, Kramarz P, van Wijk MA, van der Lei J, Sturkenboom MC. Management of hypertension and hypercholesterolaemia in primary care in The Netherlands. Curr Med Res Opin. 2005 Jun;21(6):839-48. doi: 10.1185/030079905X46368. PMID 15969884
- [Background] Nederlands Huisartsen Genootschap (NHG). NHG-standaard Cardiovasculair Risicomanagement. 2006 Jan.
- [Background] Stuurman-Bieze AG, de Boer WO, Kokenberg ME, Hugtenburg JG, de Jong-van den Berg LT, Tromp TF. Complex pharmaceutical care intervention in pulmonary care: part A. The process and pharmacists' professional satisfaction. Pharm World Sci. 2005 Oct;27(5):376-84. doi: 10.1007/s11096-005-7112-9. PMID 16341744
- [Derived] Van de Steeg-van Gompel CH, Wensing M, De Smet PA. Implementation of patient education at first and second dispensing of statins in Dutch community pharmacies: the sequel of a cluster randomized trial. BMC Health Serv Res. 2011 Nov 16;11:313. doi: 10.1186/1472-6963-11-313. PMID 22087850